CLINICAL TRIAL: NCT03036098
Title: A Phase 3, Open-label, Randomized Study of Nivolumab Combined With Ipilimumab, or With Standard of Care Chemotherapy, Versus Standard of Care Chemotherapy in Participants With Previously Untreated Unresectable or Metastatic Urothelial Cancer
Brief Title: Study of Nivolumab in Combination With Ipilimumab or Standard of Care Chemotherapy Compared to the Standard of Care Chemotherapy Alone in Treatment of Participants With Untreated Inoperable or Metastatic Urothelial Cancer
Acronym: CheckMate901
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-901; 2016-003881-14 (EudraCT Number)
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Results first posted 2025-09-18 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Urothelial Cancer
MeSH Terms: interventions — Nivolumab; Ipilimumab; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Investigational immunotherapy (Experimental)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm B: Standard of care chemotherapy (Active Comparator)
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin
- Arm C: Investigational immunotherapy (Experimental)
  Interventions: Biological: Nivolumab; Drug: Gemcitabine; Drug: Cisplatin
- Arm D: Standard of care chemotherapy (Active Comparator)
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Biological: Nivolumab — Specified Dose on Specified Days
  Other Names: BMS-936558; Opdivo
  Arms: Arm A: Investigational immunotherapy; Arm C: Investigational immunotherapy
Biological: Ipilimumab — Specified Dose on Specified Days
  Other Names: BMS-734016; Yervoy
  Arms: Arm A: Investigational immunotherapy
Drug: Gemcitabine — Specified Dose on Specified Days
  Arms: Arm B: Standard of care chemotherapy; Arm C: Investigational immunotherapy; Arm D: Standard of care chemotherapy
Drug: Cisplatin — Specified Dose on Specified Days
  Arms: Arm B: Standard of care chemotherapy; Arm C: Investigational immunotherapy; Arm D: Standard of care chemotherapy
Drug: Carboplatin — Specified Dose on Specified Days
  Arms: Arm B: Standard of care chemotherapy

SUMMARY:
The purpose of this study is to determine whether an investigational immunotherapy nivolumab in combination with ipilimumab or in combination with standard of care chemotherapy is more effective than standard of care chemotherapy alone in treating participants with previously untreated inoperable or metastatic urothelial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological evidence of metastatic or surgically inoperable transitional cell cancer (TCC) of the urothelium involving the renal pelvis, ureter, bladder or urethra
* No prior systemic chemotherapy for metastatic or surgically inoperable urothelial cancer (UC)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Women and men must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Disease that is suitable for local therapy administered with curative intent
* Any serious or uncontrolled medical disorder in the opinion of the investigator that may increase the risk associated with study participation or study drug administration or interfere with the interpretation of study results
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1314 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2026-02-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (174):
- United States (29):
  - Local Institution - 0001, Anchorage, Alaska
  - Local Institution - 0115, Fresno, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Local Institution - 0051, Boca Raton, Florida
  - Local Institution - 0087, Fort Lauderdale, Florida
  - Local Institution - 0062, Jacksonville, Florida
  - Local Institution - 0004, Athens, Georgia
  - Local Institution - 0033, Thomasville, Georgia
  - Local Institution - 0046, Chicago, Illinois
  - Local Institution - 0117, New Orleans, Louisiana
  - Local Institution - 0056, Boston, Massachusetts
  - Local Institution - 0073, Boston, Massachusetts
  - Local Institution - 0208, Boston, Massachusetts
  - Local Institution - 0207, Milford, Massachusetts
  - Local Institution - 0063, Ann Arbor, Michigan
  - Local Institution - 0002, Burnsville, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Local Institution - 0032, Kansas City, Missouri
  - Local Institution - 0095, St Louis, Missouri
  - Local Institution - 0057, Manchester, New Hampshire
  - Local Institution - 0084, Albuquerque, New Mexico
  - Local Institution - 0083, Buffalo, New York
  - Local Institution - 0014, Mineola, New York
  - Local Institution - 0072, New York, New York
  - Local Institution - 0116, Durham, North Carolina
  - Local Institution - 0082, Columbus, Ohio
  - Local Institution - 0104, Portland, Oregon
  - Local Institution - 0013, Pittsburgh, Pennsylvania
  - Local Institution - 0086, Kirkland, Washington
- Argentina (6):
  - Local Institution - 0005, Capital Federal, Buenos Aires
  - Local Institution - 0007, Mar del Plata, Buenos Aires
  - Local Institution - 0009, Buenos Aires
  - Local Institution - 0134, Córdoba
  - Local Institution - 0006, Córdoba
  - Local Institution - 0008, Viedma
- Australia (6):
  - Local Institution - 0096, Waratah, New South Wales
  - Local Institution - 0099, Westmead, New South Wales
  - Local Institution - 0188, South Brisbane, Queensland
  - Local Institution - 0120, Tugun, Queensland
  - Local Institution - 0101, Heidelberg, Victoria
  - Local Institution - 0100, Doubleview, Western Australia
- Brazil (7):
  - Local Institution - 0017, Brasília, Federal District
  - Local Institution - 0021, Ijuí, Rio Grande do Sul
  - Local Institution - 0119, Passo Fundo, Rio Grande do Sul
  - Local Institution - 0020, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0016, Florianópolis, Santa Catarina
  - Local Institution - 0018, Barretos, São Paulo
  - Local Institution - 0019, São José do Rio Preto, São Paulo
- Canada (4):
  - Local Institution - 0053, Halifax, Nova Scotia
  - Local Institution - 0064, London, Ontario
  - Local Institution - 0054, Québec, Quebec
  - Local Institution - 0052, Sherbrooke, Quebec
- Chile (3):
  - Local Institution - 0012, Viña del Mar, Región de Valparaíso
  - Local Institution - 0010, Santiago, Santiago Metropolitan
  - Local Institution - 0106, Vitacura
- China (21):
  - Local Institution - 0171, Beijing, Beijing Municipality
  - Local Institution - 0169, Beijing, Beijing Municipality
  - Local Institution - 0182, Chongqing, Chongqing Municipality
  - Local Institution - 0217, Guiyang, Guizhou
  - Local Institution - 0219, Harbin, Heilongjiang
  - Local Institution - 0180, Wuhan, Hubei
  - Local Institution - 0175, Nanjing, Jiangsu
  - Local Institution - 0177, Nanjing, Jiangsu
  - Local Institution - 0176, Nanjing, Jiangsu
  - Local Institution - 0186, Changchun, Jilin
  - Local Institution - 0220, Taiyuan, Shan1xi
  - Local Institution - 0216, Yantai, Shandong
  - Local Institution - 0167, Shanghai, Shanghai Municipality
  - Local Institution - 0162, Shanghai, Shanghai Municipality
  - Local Institution - 0163, Shanghai, Shanghai Municipality
  - Local Institution - 0184, Chengdu, Sichuan
  - Local Institution - 0173, Hangzhou, Zhejiang
  - Local Institution - 0174, Hangzhou, Zhejiang
  - Local Institution - 0172, Hangzhou, Zhejiang
  - Local Institution - 0170, Beijing
  - Local Institution - 0164, Shanghai
- Czechia (2):
  - Local Institution - 0160, Brno
  - Local Institution - 0152, Hradec Králové
- Denmark (2):
  - Local Institution - 0190, Aalborg
  - Local Institution - 0196, Herlev
- Local Institution - 0060, Helsinki, Finland
- France (7):
  - Local Institution - 0091, Nîmes, Gard
  - Local Institution - 0089, Lille
  - Local Institution - 0088, Marseille
  - Local Institution - 0090, Saint-Priest-en-Jarez
  - Local Institution - 0092, Suresnes
  - Local Institution - 0093, Tours
  - Local Institution - 0094, Villejuif
- Germany (11):
  - Local Institution - 0036, Dresden
  - Local Institution - 0048, Essen
  - Local Institution - 0047, Freiburg im Breisgau
  - Local Institution - 0049, Hamburg
  - Local Institution - 0037, Hanover
  - Local Institution - 0041, Jena
  - Local Institution - 0213, Mannheim
  - Local Institution - 0038, Nuremberg
  - Local Institution - 0040, Tübingen
  - Local Institution - 0114, Weiden
  - Local Institution - 0039, Würzburg
- Greece (2):
  - Local Institution - 0102, Athens
  - Local Institution - 0103, Ioannina, Ípeiros
- Israel (2):
  - Local Institution - 0199, Kfar Saba
  - Local Institution - 0198, Ramat Gan
- Italy (6):
  - Local Institution - 0108, Arezzo
  - Local Institution - 0197, Faenza
  - Local Institution - 0111, Forlì
  - Local Institution - 0109, Grosseto
  - Local Institution - 0107, Milan
  - Local Institution - 0110, Napoli
- Japan (20):
  - Local Institution - 0136, Hirosaki, Aomori
  - Local Institution - 0135, Chiba, Chiba
  - Local Institution - 0147, Matsuyama, Ehime
  - Local Institution - 0140, Fukuoka, Fukuoka
  - Local Institution - 0146, Sapporo, Hokkaido
  - Local Institution - 0150, Tsukuba, Ibaraki
  - Local Institution - 0214, Morioka, Iwate
  - Local Institution - 0137, Kita-Gun, Kagawa-ken
  - Local Institution - 0141, Niigata, Niigata
  - Local Institution - 0143, Okayama, Okayama-ken
  - Local Institution - 0144, Osaka, Osaka
  - Local Institution - 0139, Sayama, Osaka
  - Local Institution - 0145, Takatsuki-shi, Osaka
  - Local Institution - 0201, Hamamatasu, Shizuoka
  - Local Institution - 0149, Adachi-ku, Tokyo
  - Local Institution - 0148, Bunkyo-ku, Tokyo
  - Local Institution - 0142, Bunkyo-ku, Tokyo
  - Local Institution - 0138, Shinjuku-Ku, Tokyo
  - Local Institution - 0215, Wakayama, Wakayama
  - Local Institution - 0200, Ube, Yamaguchi
- Mexico (4):
  - Local Institution - 0129, Mexico City, Mexico City
  - Local Institution - 0154, Mexico City, Mexico City
  - Local Institution - 0130, Tlalpan, Mexico City
  - Local Institution - 0131, Monterrey, Nuevo León
- Netherlands (4):
  - Local Institution - 0022, Amsterdam, North Holland
  - Local Institution - 0055, Enschede
  - Local Institution - 0024, Groningen
  - Local Institution - 0026, Leeuwarden
- Norway (2):
  - Local Institution - 0074, Bergen
  - Local Institution - 0081, Lorenskog
- Peru (2):
  - Local Institution - 0031, Lima
  - Local Institution - 0030, Lima
- Poland (3):
  - Local Institution - 0189, Bydgoszcz
  - Local Institution - 0205, Koszalin
  - Local Institution - 0202, Warsaw
- Romania (2):
  - Local Institution - 0191, Cluj-Napoca, Cluj
  - Local Institution - 0187, Craiova, Dolj
- Local Institution, Moscow, Russia
- Local Institution - 0192, Singapore, Central Singapore, Singapore
- South Korea (6):
  - Local Institution - 0125, Goyang-si, Gyeonggido
  - Local Institution - 0126, Seongnam-si
  - Local Institution - 0124, Seoul
  - Local Institution - 0151, Seoul
  - Local Institution - 0128, Seoul
  - Local Institution - 0127, Seoul
- Spain (7):
  - Local Institution - 0070, A Coruña
  - Local Institution - 0068, Barcelona
  - Local Institution - 0065, Madrid
  - Local Institution - 0066, Madrid
  - Local Institution - 0209, Santander
  - Local Institution - 0067, Seville
  - Local Institution - 0069, Valencia
- Sweden (3):
  - Local Institution - 0075, Jönköping
  - Local Institution - 0059, Linköping
  - Local Institution - 0058, Lund
- Switzerland (2):
  - Local Institution - 0061, Baden, Canton of Aargau
  - Local Institution - 0042, Chur
- Taiwan (5):
  - Local Institution - 0156, Kaohsiung City
  - Local Institution - 0159, Taichung
  - Local Institution - 0158, Taipei
  - Local Institution - 0155, Taipei
  - Local Institution - 0157, Taoyuan District
- Turkey (Türkiye) (3):
  - Local Institution - 0194, Ankara
  - Local Institution - 0204, Istanbul
  - Local Institution - 0193, Izmir

REFERENCES:
- [Derived] Tomita Y, Ye DW, Fujii A, Takeuchi N. Nivolumab plus gemcitabine-cisplatin for previously untreated unresectable or metastatic urothelial carcinoma: an Asian subgroup analysis from the global phase 3 CheckMate 901 trial. Urol Oncol. 2025 Dec;43(12):696.e9-696.e16. doi: 10.1016/j.urolonc.2025.08.022. Epub 2025 Sep 26. PMID 41015742
- [Derived] van der Heijden MS, Sonpavde G, Powles T, Necchi A, Burotto M, Schenker M, Sade JP, Bamias A, Beuzeboc P, Bedke J, Oldenburg J, Chatta G, Urun Y, Ye D, He Z, Valderrama BP, Ku JH, Tomita Y, Filian J, Wang L, Purcea D, Patel MY, Nasroulah F, Galsky MD; CheckMate 901 Trial Investigators. Nivolumab plus Gemcitabine-Cisplatin in Advanced Urothelial Carcinoma. N Engl J Med. 2023 Nov 9;389(19):1778-1789. doi: 10.1056/NEJMoa2309863. Epub 2023 Oct 22. PMID 37870949
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT03036098.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted as a primary study and a sub-study. In the primary study, 706 participants were randomized, and 673 participants received treatment. Of these 673 treated participants, 3 were randomized in the sub-study. In the sub-study, 608 participants were randomized, and 605 participants received treatment. Of these 605 treated participants, 13 were randomized in the primary study.
Groups:
- Treatment 1: Participants received Nivolumab 1 mg/kg plus Ipilimumab 3 mg/kg every three weeks (Q3W) for up to 4 doses followed by Nivolumab monotherapy 480 mg every 4 weeks (Q4W) - Primary Study
- Treatment 2: Participants received Standard of Care treatment every three weeks (Q3W) for up to 6 cycles - Primary Study
- Treatment 3: Participants received Nivolumab 360 mg in combination with Standard of Care treatment every 3 weeks (Q3W) for up to 6 cycles followed by Nivolumab monotherapy 480 mg every 4 weeks (Q4W) - Sub-study
- Treatment 4: Participants received Standard of Care treatment every three weeks (Q3W) for up to 6 cycles - Sub-study
Period: Pre-Treatment
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Started (Started = Randomized) | 349 | 357 | 304 | 304
Completed (Completed = Treated) | 345 | 338 (13 participants were randomized to Treatment 2; however, they received the sub-study treatment (Treatment 4)) | 304 | 291 (3 participants were randomized to Treatment 4; however, they received the primary study treatment (Treatment 2))
Not Completed | 4 | 19 | 0 | 13
Not completed — Other Reasons | 1 | 2 | 0 | 5
Not completed — Participant No Longer Meets Study Criteria | 2 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 14 | 0 | 5
Not completed — Participant Request to Discontinue Study Treatment | 0 | 3 | 0 | 1
Period: Treatment
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Started (Started = Treated) | 345 | 325 | 304 | 288
Received Different Treatment Than Originally Assigned | 0 | 13 (13 participants were randomized in primary study (Treatment 2); however, they received the sub-study treatment (Treatment 4)) | 0 | 3 (3 participants were randomized in sub-study (Treatment 4); however, they received the primary study treatment (Treatment 2))
Completed | 46 | 149 | 29 | 157
Not Completed | 299 | 176 | 275 | 131
Not completed — Disease Progression | 130 | 77 | 168 | 50
Not completed — Study Drug Toxicity | 95 | 45 | 26 | 22
Not completed — Death | 9 | 3 | 1 | 2
Not completed — Adverse Event Unrelated to Study Drug | 18 | 15 | 10 | 14
Not completed — Participant Request to Discontinue Study Treatment | 6 | 18 | 15 | 18
Not completed — Withdrawal by Subject | 2 | 9 | 2 | 4
Not completed — Maximum Clinical Benefit | 6 | 1 | 6 | 10
Not completed — Poor/Non Compliance | 1 | 2 | 0 | 1
Not completed — Participant No Longer Meets Study Criteria | 0 | 1 | 1 | 1
Not completed — Administrative Reason by Sponsor | 1 | 0 | 2 | 1
Not completed — Other Reasons | 31 | 5 | 21 | 8
Not completed — Ongoing Treatment | 0 | 0 | 23 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Total
Number analyzed (Participants) | 349 | 357 | 304 | 304 | 1314
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 120 | 127 | 150 | 148 | 545
  >=65 years | 229 | 230 | 154 | 156 | 769
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 88 | 68 | 70 | 306
  Male | 269 | 269 | 236 | 234 | 1008
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 18 | 38 | 33 | 113
  Not Hispanic or Latino | 158 | 151 | 118 | 119 | 546
  Unknown or Not Reported | 167 | 188 | 148 | 152 | 655
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 253 | 232 | 211 | 225 | 921
  Black Or African American | 1 | 1 | 0 | 2 | 4
  American Indian Or Alaska Native | 2 | 2 | 1 | 1 | 6
  Asian | 79 | 105 | 75 | 63 | 322
  Other | 14 | 16 | 17 | 13 | 60
  Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Cisplatin-ineligible Randomized Participants for Primary Study
Description: This measure looks at how long participants who cannot receive cisplatin (a type of chemotherapy) live after being placed into a treatment group in the primary study.
  Overall Survival (OS) is defined as the time between the date a participant is randomized (assigned to a treatment group) and the date of death from any cause. For participants without documentation of death, OS will be measured up to the last date the participant was known to be alive. If a participant was randomized but had no follow-up information, OS will be counted from the date of randomization.
  This helps to understand if the treatment can help people who are unable to receive cisplatin chemotherapy live longer.
Time Frame: From the date of randomization to the date of death from any cause, or data cut-off date, whichever occurred first (up to approximately 89 months)
Population: All Cisplatin-ineligible Randomized Participants - Primary Study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 221 | 224
Months | 19.06 [13.47 to 22.60] | 13.21 [11.63 to 15.24]
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; Test type: Superiority; p = 0.0032, Log Rank; Stratified weighted log-rank test; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.64 to 0.97]

2. Primary Outcome: Overall Survival (OS) in Programmed Death-Ligand 1 (PD-L1) Positive (≥ 1%) Randomized Participants by Immunohistochemistry (IHC) for Primary Study
Description: This measure looks at how long participants with PD-L1 positive tumors (meaning their tumor cells have at least 1% PD-L1, as determined by a laboratory test called immunohistochemistry or IHC) live after being placed into a treatment group in the primary study.
  Overall Survival (OS) is defined as the time between the date a participant is randomized (assigned to a treatment group) and the date of death from any cause. For participants without documentation of death, OS will be measured up to the last date the participant was known to be alive. If a participant was randomized but had no follow-up information, OS will be counted from the date of randomization.
  This helps to understand whether the treatment can help people with PD-L1 positive tumors live longer.
Time Frame: as for outcome 1
Population: All PD-L1 >= 1% Randomized Participants - Primary Study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 123 | 127
Months | 16.30 [11.53 to 21.82] | 14.36 [10.48 to 17.64]

3. Secondary Outcome: Overall Survival (OS) in All Randomized Participants for Primary Study
Description: This measure looks at how long all participants live after being placed into a treatment group in the primary study.
  Overall Survival (OS) is defined as the time between the date a participant is randomized (assigned to a treatment group) and the date of death from any cause. For participants without documentation of death, OS will be measured up to the last date the participant was known to be alive. If a participant was randomized but had no follow-up information, OS will be counted from the date of randomization.
  This helps to understand whether the treatment can help all participants in the study live longer.
Time Frame: as for outcome 1
Population: All Randomized Participants - Primary Study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 349 | 357
Months | 18.76 [15.05 to 21.82] | 14.32 [12.22 to 15.87]

4. Secondary Outcome: Progression-Free Survival (PFS) by Blinded Independent Central Review (BICR) [Using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1] in Cisplatin-ineligible Randomized Participants for Primary Study
Description: This measure looks at how long people who cannot receive cisplatin chemotherapy live without their cancer getting worse after being assigned to a treatment group in the primary study. Progression-Free Survival (PFS) is the time from when a participant is assigned to a group (randomization) until their cancer is first shown to get worse (progress), based on reviews by independent experts who do not know which treatment was given. These experts use standard rules (RECIST 1.1) to decide if the cancer has progressed. If a participant dies before their cancer is shown to get worse, the date of death will be used as the time their disease progressed. If a participant's cancer does not get worse and they do not die during the study, their PFS will be measured up to the date of their last tumor check. This helps to understand if the treatment helps people unable to receive cisplatin live longer without their cancer progressing.
Time Frame: From the date of randomization to the date of first documented disease progression or death due to any cause, whichever occurs first (up to approximately 89 months)
Population: All Cisplatin-ineligible Randomized Participants - Primary Study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 221 | 224
Months | 5.29 [3.78 to 5.95] | 5.88 [5.62 to 7.59]

5. Secondary Outcome: Progression-Free Survival (PFS) by Blinded Independent Central Review (BICR) [Using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1] in Programmed Death-Ligand 1 (PD-L1) Positive (≥ 1%) Participants for Primary Study
Description: This measure looks at how long people with PD-L1 positive tumors (meaning their tumor cells have at least 1% PD-L1, as determined by a lab test) live without their cancer getting worse after being assigned to a treatment group in the primary study. Progression-Free Survival (PFS) is the time from when a participant is assigned to a group (randomization) until their cancer is first shown to get worse (progress), based on reviews by independent experts who do not know which treatment was given. These experts use standard rules (RECIST 1.1) to decide if the cancer has progressed. If a participant dies before their cancer is shown to get worse, the date of death will be used as the time their disease progressed. If a participant's cancer does not get worse and they do not die during the study, their PFS will be measured up to the date of their last tumor check. This helps to understand if the treatment helps people with PD-L1 positive tumors live longer without their cancer progressing.
Time Frame: as for outcome 4
Population: All PD-L1 >= 1% Randomized Participants - Primary Study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 123 | 127
Months | 5.39 [3.75 to 7.39] | 5.78 [4.80 to 6.93]

6. Secondary Outcome: Progression-Free Survival (PFS) by Blinded Independent Central Review (BICR) [Using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1] in All Randomized Participants for Primary Study
Description: This measure looks at how long all participants in the primary study live without their cancer getting worse after being assigned to a treatment group.
  Progression-Free Survival (PFS) is defined as the time from when a participant is assigned to a treatment group (randomization) until their cancer is first shown to get worse (progress), based on reviews by independent experts who do not know which treatment the participant received. These experts use standard rules (called RECIST 1.1) to decide if the cancer has progressed. If a participant dies before their cancer is shown to get worse, the date of death will be used as the time their disease progressed. If a participant's cancer does not get worse and they do not die during the study, their PFS will be measured up to the date of their last tumor check.
  This helps to understand whether the treatment can help participants live longer without their cancer progressing.
Time Frame: as for outcome 4
Population: All Randomized Participants - Primary Study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 349 | 357
Months | 5.03 [3.94 to 5.98] | 6.01 [5.78 to 7.52]

7. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Care Quality-of-Life Questionnaire (EORTC QLQ-C30) Global Health Status Score in All Randomized Participants for Primary Study
Description: The EORTC QLQ-C30 is a questionnaire used to assess the quality of life in cancer patients. It includes a global health status score, which is measured on a 4-point Likert scale: 1 = not at all, 2 = a little, 3 = quite a bit, and 4 = very much. Responses are combined and converted to scores ranging from 0 to 100. A high score for global health status or health-related quality of life (HRQoL) indicates a high overall HRQoL.
Time Frame: At Baseline, Week 4, Week 10, Week 16, Week 20, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96, Week 108, Week 120, Week 144, Week 156, Week 168, Week 180 and Week 192
Population: All Randomized Participants - Primary Study
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 349 | 357
Score on a Scale
  Global Health Status - Baseline: number analyzed (Participants) | 322 | 316
  Global Health Status - Baseline | 63.4 (22.55) | 59.8 (25.05)
  Global Health Status - Week 4: number analyzed (Participants) | 244 | 249
  Global Health Status - Week 4 | -1.1 (18.28) | 2.7 (23.21)
  Global Health Status - Week 10: number analyzed (Participants) | 159 | 204
  Global Health Status - Week 10 | -0.5 (23.73) | 3.0 (23.55)
  Global Health Status - Week 16: number analyzed (Participants) | 117 | 132
  Global Health Status - Week 16 | 3.6 (22.59) | 3.1 (24.68)
  Global Health Status - Week 20: number analyzed (Participants) | 103 | 67
  Global Health Status - Week 20 | 2.6 (22.02) | 5.1 (24.44)
  Global Health Status - Week 24: number analyzed (Participants) | 106 | 36
  Global Health Status - Week 24 | 1.9 (25.78) | 2.5 (26.19)
  Global Health Status - Week 36: number analyzed (Participants) | 89 | 10
  Global Health Status - Week 36 | -0.9 (22.14) | -1.7 (28.81)
  Global Health Status - Week 48: number analyzed (Participants) | 62 | 3
  Global Health Status - Week 48 | 0.5 (19.72) | 2.8 (17.35)
  Global Health Status - Week 60: number analyzed (Participants) | 56 | 0
  Global Health Status - Week 60 | 7.6 (24.11) |
  Global Health Status - Week 72: number analyzed (Participants) | 47 | 0
  Global Health Status - Week 72 | 2.7 (27.04) |
  Global Health Status - Week 84: number analyzed (Participants) | 34 | 0
  Global Health Status - Week 84 | 8.1 (24.40) |
  Global Health Status - Week 96: number analyzed (Participants) | 29 | 0
  Global Health Status - Week 96 | 3.2 (26.86) |
  Global Health Status - Week 108: number analyzed (Participants) | 16 | 0
  Global Health Status - Week 108 | 4.7 (37.51) |
  Global Health Status - Week 120: number analyzed (Participants) | 4 | 0
  Global Health Status - Week 120 | -20.8 (28.46) |
  Global Health Status - Week 144: number analyzed (Participants) | 1 | 0
  Global Health Status - Week 144 | -16.7 (NA) — Insufficient number of participants to calculate SD. |
  Global Health Status - Week 156: number analyzed (Participants) | 1 | 0
  Global Health Status - Week 156 | -16.7 (NA) — Insufficient number of participants to calculate SD. |
  Global Health Status - Week 168: number analyzed (Participants) | 1 | 0
  Global Health Status - Week 168 | 0.0 (NA) — Insufficient number of participants to calculate SD. |
  Global Health Status - Week 180: number analyzed (Participants) | 1 | 0
  Global Health Status - Week 180 | -8.3 (NA) — Insufficient number of participants to calculate SD. |
  Global Health Status - Week 192: number analyzed (Participants) | 1 | 0
  Global Health Status - Week 192 | -16.7 (NA) — Insufficient number of participants to calculate SD. |

8. Primary Outcome: Progression-Free Survival (PFS) by Blinded Independent Central Review (BICR) [Using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1] in Cisplatin-eligible Participants for Sub-study
Description: This measure looks at how long people who can receive cisplatin chemotherapy live without their cancer getting worse after being assigned to a treatment group in the sub-study. Progression-Free Survival (PFS) is the time from when a participant is assigned to a group (randomization) until their cancer is first shown to get worse (progress), based on reviews by independent experts who do not know which treatment was given. These experts use standard rules (RECIST 1.1) to decide if the cancer has progressed. If a participant dies before their cancer is shown to get worse, the date of death will be used as the time their disease progressed. If a participant's cancer does not get worse and they do not die during the study, their PFS will be measured up to the date of their last tumor check. This helps to understand if the treatment helps people eligible for cisplatin live longer without their cancer progressing.
Time Frame: as for outcome 4
Population: All Cisplatin-eligible Randomized Participants - Sub-study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 3 | Treatment 4
Number analyzed (Participants) | 304 | 304
Months | 7.92 [7.62 to 9.49] | 7.56 [6.05 to 7.75]
Statistical Analysis 1: Comparison: Treatment 3 vs Treatment 4; Test type: Superiority; p = 0.0018, Log Rank; Stratified weighted log-rank test; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.59 to 0.88]

9. Primary Outcome: Overall Survival (OS) in Cisplatin-eligible Participants for Sub-study
Description: This measure looks at how long people who are able to receive cisplatin (a type of chemotherapy) live after being placed into a treatment group in the sub-study.
  Overall Survival (OS) is defined as the time between the date a participant is randomized (assigned to a treatment group) and the date of death from any cause. For participants without documentation of death, OS will be measured up to the last date the participant was known to be alive. If a participant was randomized but had no follow-up information, OS will be counted from the date of randomization.
  This helps to understand if the treatment can help people who are eligible for cisplatin chemotherapy live longer.
Time Frame: as for outcome 1
Population: All Cisplatin-eligible Randomized Participants - Sub-study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 3 | Treatment 4
Number analyzed (Participants) | 304 | 304
Months | 21.72 [18.63 to 26.38] | 18.86 [14.72 to 22.44]
Statistical Analysis 1: Comparison: Treatment 3 vs Treatment 4; Test type: Superiority; p = 0.0171, Log Rank; Stratified weighted log-rank test; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.63 to 0.96]

10. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Care Quality-of-Life Questionnaire (EORTC QLQ-C30) Global Health Status Score for Sub-study
Description: as for outcome 7
Time Frame: At Baseline, Week 4, Week 10, Week 16, Week 20, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96, Week 108, and Week 120
Population: All Randomized Participants - Sub-study
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Treatment 3 | Treatment 4
Number analyzed (Participants) | 304 | 304
Score on a Scale
  Global Health Status - Baseline: number analyzed (Participants) | 291 | 274
  Global Health Status - Baseline | 66.6 (22.7) | 66.8 (22.5)
  Global Health Status - Week 4: number analyzed (Participants) | 245 | 218
  Global Health Status - Week 4 | -0.2 (22.2) | 2.0 (17.8)
  Global Health Status - Week 10: number analyzed (Participants) | 238 | 187
  Global Health Status - Week 10 | 2.9 (24.2) | 1.1 (20.6)
  Global Health Status - Week 16: number analyzed (Participants) | 106 | 135
  Global Health Status - Week 16 | 1.8 (23.1) | -1.0 (23.7)
  Global Health Status - Week 20: number analyzed (Participants) | 165 | 50
  Global Health Status - Week 20 | 4.3 (24.6) | -0.5 (22.8)
  Global Health Status - Week 24: number analyzed (Participants) | 193 | 29
  Global Health Status - Week 24 | 4.0 (25.3) | -0.6 (13.0)
  Global Health Status - Week 36: number analyzed (Participants) | 150 | 9
  Global Health Status - Week 36 | 6.4 (25.1) | -3.7 (17.2)
  Global Health Status - Week 48: number analyzed (Participants) | 92 | 3
  Global Health Status - Week 48 | 7.1 (24.9) | -2.8 (12.7)
  Global Health Status - Week 60: number analyzed (Participants) | 62 | 0
  Global Health Status - Week 60 | 8.1 (25.0) |
  Global Health Status - Week 72: number analyzed (Participants) | 54 | 1
  Global Health Status - Week 72 | 6.6 (26.5) | -8.3 (NA) — Insufficient number of participants to calculate SD.
  Global Health Status - Week 84: number analyzed (Participants) | 39 | 0
  Global Health Status - Week 84 | 9.8 (26.7) |
  Global Health Status - Week 96: number analyzed (Participants) | 26 | 0
  Global Health Status - Week 96 | 9.0 (18.2) |
  Global Health Status - Week 108: number analyzed (Participants) | 11 | 0
  Global Health Status - Week 108 | 7.6 (13.7) |
  Global Health Status - Week 120: number analyzed (Participants) | 3 | 0
  Global Health Status - Week 120 | 13.9 (25.5) |

11. Secondary Outcome: Progression-Free Survival (PFS) by Blinded Independent Central Review (BICR) [Using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1] by Programmed Death-Ligand 1 (PD-L1) Expression at ≥1% Expression by Immunohistochemistry (IHC) for Sub-study
Description: This measure looks at how long participants with PD-L1 positive tumors (meaning their tumor cells have at least 1% PD-L1, as determined by a lab test called immunohistochemistry or IHC) live without their cancer getting worse after being assigned to a treatment group in the sub-study.
  Progression-Free Survival (PFS) is the time from when a participant is assigned to a group (randomization) until their cancer is first shown to get worse (progress), based on reviews by independent experts who do not know which treatment was given. These experts use standard rules (RECIST 1.1) to decide if the cancer has progressed. If a participant dies before their cancer is shown to get worse, the date of death will be used as the time their disease progressed. If a participant's cancer does not get worse and they do not die during the study, their PFS will be measured up to the date of their last tumor check.
Time Frame: as for outcome 4
Population: All PD-L1 >= 1% Randomized Participants - Sub-study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 3 | Treatment 4
Number analyzed (Participants) | 111 | 110
Months | 8.08 [7.10 to 11.27] | 6.60 [5.78 to 7.59]

12. Secondary Outcome: Overall Survival (OS) by Blinded Independent Central Review (BICR) [Using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1] by Programmed Death-Ligand 1 (PD-L1) Expression at ≥1% Expression by Immunohistochemistry (IHC) for Sub-study
Description: This measure looks at how long participants with PD-L1 positive tumors (meaning their tumor cells have at least 1% PD-L1, as determined by a laboratory test called immunohistochemistry or IHC) live after being placed into a treatment group in the sub-study.
  Overall Survival (OS) is defined as the time between the date a participant is randomized (assigned to a treatment group) and the date of death from any cause. For participants without documentation of death, OS will be measured up to the last date the participant was known to be alive. If a participant was randomized but had no follow-up information, OS will be counted from the date of randomization.
  This helps to understand whether the treatment can help people with PD-L1 positive tumors live longer. The results are reviewed by independent experts who do not know which treatment each participant received, using standard criteria for measuring tumor response.
Time Frame: as for outcome 1
Population: All PD-L1 >= 1% Randomized Participants - Sub-study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 3 | Treatment 4
Number analyzed (Participants) | 111 | 110
Months | 25.10 [17.28 to 35.55] | 15.34 [11.70 to 24.87]

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from the date of randomization until primary study completion. SAEs and Other AEs were assessed from first dose of study medication until primary study completion (assessed up to approximately 89 months).
Description: All-Cause Mortality represents all randomized participants. Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
All-Cause Mortality (participants affected / at risk) | 257/349 | 294/357 | 172/304 | 193/304
Serious Adverse Events (participants affected / at risk) | 264/345 | 170/328 | 168/304 | 130/301
Other Adverse Events (participants affected / at risk) | 322/345 | 309/328 | 298/304 | 295/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=345) | Treatment 2 (N=328) | Treatment 3 (N=304) | Treatment 4 (N=301)
Anaemia (Blood and lymphatic system disorders) | 6 | 18 | 9 | 8
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Bicytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Cytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 4 | 2
Immune-mediated pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 0 | 4 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 10 | 6 | 3
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 1 | 0
Autoimmune myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 1
Immune-mediated myocarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2 | 0 | 1
Myocardial injury (Cardiac disorders) | 0 | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 3 | 0 | 2 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 10 | 0 | 1 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0 | 0 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 | 0 | 1 | 0
Glucocorticoid deficiency (Endocrine disorders) | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 3 | 0 | 1 | 0
Hypophysitis (Endocrine disorders) | 8 | 0 | 1 | 0
Hypopituitarism (Endocrine disorders) | 3 | 0 | 2 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0 | 0 | 0
Immune-mediated hypophysitis (Endocrine disorders) | 1 | 0 | 0 | 0
Immune-mediated thyroiditis (Endocrine disorders) | 1 | 0 | 0 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 2 | 0 | 0 | 0
Age-related macular degeneration (Eye disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 2 | 0
Papilloedema (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Autoimmune colitis (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Autoimmune enteropathy (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 16 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 19 | 2 | 1 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 9 | 0 | 2 | 0
Immune-mediated pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 6 | 6 | 2
Intestinal perforation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Oesophageal rupture (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 1 | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Rectal lesion (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1 | 3 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 4 | 3
Asthenia (General disorders) | 1 | 1 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 2 | 0 | 0 | 0
Device related thrombosis (General disorders) | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 3 | 0 | 1 | 1
General physical health deterioration (General disorders) | 3 | 2 | 4 | 2
Hyperpyrexia (General disorders) | 2 | 0 | 0 | 0
Hyperthermia (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 3 | 0 | 0 | 3
Multiple organ dysfunction syndrome (General disorders) | 1 | 3 | 2 | 2
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1
Pain (General disorders) | 5 | 2 | 0 | 3
Pelvic mass (General disorders) | 0 | 1 | 0 | 0
Performance status decreased (General disorders) | 0 | 1 | 0 | 0
Polyserositis (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 13 | 9 | 6 | 4
Sudden death (General disorders) | 7 | 4 | 1 | 2
Systemic inflammatory response syndrome (General disorders) | 2 | 0 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 2 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 5 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 3 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 12 | 0 | 1 | 0
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Suspected drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Abdominal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Aeromonas infection (Infections and infestations) | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 6 | 3
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Clostridium colitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 1 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 0 | 0 | 0
Device related bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 2 | 2 | 2 | 2
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1 | 0
Empyema (Infections and infestations) | 1 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 2 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 1
Epiglottitis (Infections and infestations) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 2 | 1 | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster meningoencephalitis (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 1 | 3 | 1
Influenza (Infections and infestations) | 2 | 0 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 2 | 0
Klebsiella urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 2 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 8 | 7 | 6 | 8
Pneumonia aspiration (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 2
Pneumonia legionella (Infections and infestations) | 1 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 2 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 3 | 4 | 2
Pyelonephritis acute (Infections and infestations) | 2 | 0 | 2 | 2
Pyonephrosis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 11 | 7 | 7 | 4
Septic shock (Infections and infestations) | 1 | 1 | 4 | 3
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 0 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
Systemic infection (Infections and infestations) | 0 | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 33 | 19 | 15 | 16
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 5 | 4 | 5 | 3
Vascular device infection (Infections and infestations) | 0 | 1 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Bladder injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Depressed fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Urostomy complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 5 | 4 | 1 | 1
General physical condition abnormal (Investigations) | 1 | 1 | 0 | 1
Heart rate irregular (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 2 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 2 | 1 | 0
Platelet count decreased (Investigations) | 0 | 12 | 7 | 1
Transaminases increased (Investigations) | 5 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 0 | 2 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 51 | 38 | 47 | 22
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 4 | 2 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 1 | 0
Encephalitis autoimmune (Nervous system disorders) | 0 | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Immune-mediated encephalitis (Nervous system disorders) | 1 | 0 | 0 | 0
Immune-mediated encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 1 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0 | 0 | 0
Neurological decompensation (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 0 | 0
Stroke in evolution (Nervous system disorders) | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 2 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 0 | 1
Device malfunction (Product Issues) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 19 | 4 | 13 | 5
Anuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Bladder stenosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Bladder tamponade (Renal and urinary disorders) | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 8 | 2 | 5 | 6
Hydronephrosis (Renal and urinary disorders) | 1 | 4 | 2 | 2
Hydroureter (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1
Postrenal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 5 | 0 | 2 | 3
Renal impairment (Renal and urinary disorders) | 0 | 1 | 2 | 0
Ureteric dilatation (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 2 | 0
Urethral disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary tract inflammation (Renal and urinary disorders) | 2 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 1 | 1
Vesicocutaneous fistula (Renal and urinary disorders) | 1 | 0 | 0 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Scrotal mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 11 | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 8 | 6
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 2 | 2
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 2 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 2 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0
Iliac vein occlusion (Vascular disorders) | 0 | 0 | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral embolism (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=345) | Treatment 2 (N=328) | Treatment 3 (N=304) | Treatment 4 (N=301)
Anaemia (Blood and lymphatic system disorders) | 82 | 195 | 193 | 170
Leukopenia (Blood and lymphatic system disorders) | 1 | 24 | 42 | 33
Neutropenia (Blood and lymphatic system disorders) | 1 | 104 | 104 | 94
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 71 | 52 | 38
Tinnitus (Ear and labyrinth disorders) | 2 | 13 | 19 | 21
Hyperthyroidism (Endocrine disorders) | 48 | 0 | 22 | 0
Hypothyroidism (Endocrine disorders) | 53 | 0 | 41 | 0
Abdominal pain (Gastrointestinal disorders) | 23 | 18 | 25 | 18
Constipation (Gastrointestinal disorders) | 53 | 90 | 92 | 86
Diarrhoea (Gastrointestinal disorders) | 113 | 46 | 59 | 46
Dyspepsia (Gastrointestinal disorders) | 9 | 19 | 14 | 10
Nausea (Gastrointestinal disorders) | 74 | 122 | 159 | 161
Vomiting (Gastrointestinal disorders) | 53 | 62 | 69 | 60
Asthenia (General disorders) | 65 | 63 | 68 | 63
Fatigue (General disorders) | 78 | 76 | 87 | 84
Malaise (General disorders) | 12 | 21 | 19 | 10
Oedema peripheral (General disorders) | 47 | 38 | 44 | 28
Pyrexia (General disorders) | 81 | 55 | 40 | 39
COVID-19 (Infections and infestations) | 2 | 0 | 19 | 5
Urinary tract infection (Infections and infestations) | 69 | 44 | 40 | 42
Alanine aminotransferase increased (Investigations) | 43 | 17 | 32 | 17
Amylase increased (Investigations) | 15 | 11 | 34 | 16
Aspartate aminotransferase increased (Investigations) | 33 | 16 | 30 | 16
Blood alkaline phosphatase increased (Investigations) | 20 | 13 | 14 | 12
Blood creatinine increased (Investigations) | 54 | 34 | 64 | 55
Lipase increased (Investigations) | 24 | 6 | 30 | 13
Lymphocyte count decreased (Investigations) | 2 | 12 | 16 | 12
Neutrophil count decreased (Investigations) | 3 | 90 | 78 | 61
Platelet count decreased (Investigations) | 7 | 76 | 67 | 50
Weight decreased (Investigations) | 36 | 14 | 33 | 18
White blood cell count decreased (Investigations) | 2 | 55 | 64 | 42
Decreased appetite (Metabolism and nutrition disorders) | 79 | 66 | 94 | 61
Hyperglycaemia (Metabolism and nutrition disorders) | 26 | 15 | 20 | 15
Hyperkalaemia (Metabolism and nutrition disorders) | 13 | 20 | 11 | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 29 | 15 | 15 | 16
Hypokalaemia (Metabolism and nutrition disorders) | 27 | 9 | 23 | 18
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 21 | 21 | 34
Hyponatraemia (Metabolism and nutrition disorders) | 30 | 15 | 36 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 | 17 | 34 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 26 | 39 | 31
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 9 | 17 | 6
Dizziness (Nervous system disorders) | 15 | 25 | 24 | 18
Dysgeusia (Nervous system disorders) | 9 | 17 | 22 | 13
Headache (Nervous system disorders) | 23 | 23 | 31 | 17
Neuropathy peripheral (Nervous system disorders) | 6 | 14 | 23 | 17
Paraesthesia (Nervous system disorders) | 5 | 4 | 16 | 17
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 8 | 16 | 9
Insomnia (Psychiatric disorders) | 30 | 24 | 19 | 16
Acute kidney injury (Renal and urinary disorders) | 19 | 5 | 13 | 15
Haematuria (Renal and urinary disorders) | 24 | 22 | 31 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 29 | 26 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 | 27 | 21 | 15
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 13 | 18 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 33 | 22 | 28
Pruritus (Skin and subcutaneous tissue disorders) | 104 | 16 | 54 | 10
Rash (Skin and subcutaneous tissue disorders) | 76 | 28 | 52 | 16
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 32 | 4 | 7 | 2
Hypertension (Vascular disorders) | 13 | 13 | 25 | 12
Hypotension (Vascular disorders) | 16 | 0 | 18 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT03036098/Prot_SAP_000.pdf